CLINICAL TRIAL: NCT04125940
Title: Blood Nitrate/Nitrite Concentrations Following Acute Ingestion of Resync in Men and Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Memphis (Other)
Collaborators: Resync, LLC (Unknown)
Responsible Party: Principal Investigator, Richard Bloomer, Dean of School of Health Studies, University of Memphis
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: PRO-FY2020-67
Record Dates: First submitted 2019-10-08; First posted 2019-10-14 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Healthy
Keywords: Resync; Nitrate; Nitrite; Healthy
MeSH Terms: interventions — Collagen

STUDY DESIGN:
Intervention Model Description: Single-blind, pre-post ingestion, control
Who Masked: Participant
Masking Description: Single-Blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo-controlled Arm (Placebo Comparator): Placebo - 12oz water with food coloring
  Interventions: Other: Placebo
- 1 serving Resync Arm (Active Comparator): 12oz water + 7.5g Resync
  Interventions: Dietary Supplement: Resync
- 2 servings Resync Arm (Active Comparator): 12oz water + 15g Resync
  Interventions: Dietary Supplement: Resync
- 1 servings Resync+Collagen Arm (Active Comparator): 12oz water + 17g collagen + 2g Resync + 1g Carbohydrates
  Interventions: Dietary Supplement: Resync + Collagen

INTERVENTIONS:
Dietary Supplement: Resync — The product known as Resync contains a blend of nitrate-rich foods including beetroot, red spinach, turmeric, ginger root, and aronia berry extracts. Resync is sold commercially and marketed as an ergogenic aid and/or exercise recovery aid.
  Arms: 1 serving Resync Arm; 2 servings Resync Arm
Dietary Supplement: Resync + Collagen — 17g Collagen + 2g Resync + 1g Carbohydrate
  Arms: 1 servings Resync+Collagen Arm
Other: Placebo — 12oz water + food coloring
  Arms: Placebo-controlled Arm

SUMMARY:
This study evaluates acute ingestion of the dietary supplement Resync on blood nitrate/nitrite concentrations in a sample of men and women. This will be a crossover trial in which participants take all 4 conditions: 1) 7.5g Resync, 2) 15g Resync, 3) 20g Resync+collagen, 4) placebo.

DETAILED DESCRIPTION:
The product known as Resync contains a blend of nitrate-rich foods including beetroot, red spinach, turmeric, ginger root, and aronia berry extracts. Resync is sold commercially and marketed as an ergogenic aid and/or exercise recovery aid. Manufacturers of Resync recommend users take this product 60-90 minutes before an athletic event or 30-90 minutes after exercise. Resync bases these claims on prior studies investigating the individual ingredients' abilities to increase blood nitrate/nitrite levels; however, there are no clinical trials on the finished product itself.

The purpose of this pilot study is to determine the impact of acute, single ingestion of Resync products on blood nitrate/nitrite concentration in a sample of men and women. This will be a crossover trial in which participants take all 4 conditions: 1) 7.5g Resync, 2) 15g Resync, 3) 20g Resync+collagen, 4) placebo.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18 - 29.9 kg/m2
* Non-smoker
* Non-vegan
* Not using nitrate-based dietary supplements

Exclusion Criteria:

* Diagnosed history of diabetes
* Diagnosed history of cardiovascular disease
* Diagnosed history of neurological disease
* Pregnant females

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Change in blood nitrate+nitrite levels from daily baseline with 7.5g Resync | 75-minutes post supplement ingestion
  We will determine the change in daily blood nitrate+nitrite from the daily baseline blood nitrate+nitrite with 1 serving (7.5g) of Resync. Resync powder will be mixed with 12oz of water.
Change in blood nitrate+nitrite levels from daily baseline with 15g Resync | 75-minutes post supplement ingestion
  We will determine the change in daily blood nitrate+nitrite from the daily baseline blood nitrate+nitrite with 2 servings (15g) of Resync. Resync powder will be mixed with 12oz of water.
Change in blood nitrate+nitrite levels from daily baseline with 20g Resync+Collagen | 75-minutes post supplement ingestion
  We will determine the change in daily blood nitrate+nitrite from the daily baseline blood nitrate+nitrite with 1 serving (20g) of Resync+Collagen. This blend contains approximately 17g of collagen, 2 g of Resync, and 1g carbohydrates. Resync+Collagen powder will be mixed with 12oz of water.
Change in blood nitrate+nitrite levels from daily baseline with placebo. | 75-minutes post supplement ingestion
  We will determine the change in daily blood nitrate+nitrite from the daily baseline blood nitrate+nitrite with 12oz of food colored water. A red food dye will be used to match coloring of supplements.
Change in systolic blood pressure from daily baseline with 7.5g Resync | 75-minutes post supplement ingestion
  We will determine the change in daily systolic blood pressure with supplementation from the daily baseline systolic blood pressure with 1 serving (7.5g) of Resync. Resync powder will be mixed with 12oz of water.
Change in systolic blood pressure from daily baseline with 15g Resync | 75-minutes post supplement ingestion
  We will determine the change in daily systolic blood pressure with supplementation from the daily baseline systolic blood pressure with 2 servings (15g) of Resync. Resync powder will be mixed with 12oz of water.
Change in systolic blood pressure from daily baseline with 20g Resync+Collagen | 75-minutes post supplement ingestion
  We will determine the change in daily systolic blood pressure with supplementation from the daily baseline systolic blood pressure with 1 serving (20g) of Resync+Collagen. This blend contains approximately 17g of collagen, 2 g of Resync, and 1g carbohydrates. Resync+Collagen powder will be mixed with 12oz of water.
Change in systolic blood pressure from daily baseline with placebo | 75-minutes post supplement ingestion
  We will determine the change in daily systolic blood pressure with supplementation from the daily baseline systolic blood pressure with 12oz of food colored water. A red food dye will be used to match coloring of supplements.
Change in diastolic blood pressure from daily baseline with 7.5g Resync | 75-minutes post supplement ingestion
  We will determine the change in daily diastolic blood pressure with supplementation from the daily baseline diastolic blood pressure with 1 serving (7.5g) of Resync. Resync powder will be mixed with 12oz of water.
Change in diastolic blood pressure from daily baseline with 15g Resync | 75-minutes post supplement ingestion
  We will determine the change in daily diastolic blood pressure with supplementation from the daily baseline diastolic blood pressure with 2 servings (15g) of Resync. Resync powder will be mixed with 12oz of water.
Change in diastolic blood pressure from daily baseline with 20g Resync+Collagen | 75-minutes post supplement ingestion
  We will determine the change in daily diastolic blood pressure with supplementation from the daily baseline diastolic blood pressure with 1 serving (20g) of Resync+Collagen. This blend contains approximately 17g of collagen, 2 g of Resync, and 1g carbohydrates. Resync+Collagen powder will be mixed with 12oz of water.
Change in diastolic blood pressure from daily baseline with placebo | 75-minutes post supplement ingestion
  We will determine the change in daily diastolic blood pressure with supplementation from the daily baseline diastolic blood pressure with 12oz of food colored water. A red food dye will be used to match coloring of supplements.

SECONDARY OUTCOMES:
Change in heart rate from daily baseline with 7.5g Resync | 75-minutes post supplement ingestion
  We will determine the change in daily heart rate with supplementation from the daily baseline heart rate with 1 serving (7.5g) of Resync. Resync powder will be mixed with 12oz of water.
Change in heart rate from daily baseline with 15g Resync | 75-minutes post supplement ingestion
  We will determine the change in daily heart rate with supplementation from the daily baseline heart rate with 2 servings (15g) of Resync. Resync powder will be mixed with 12oz of water.
Change in heart rate from daily baseline with placebo | 75-minutes post supplement ingestion
  We will determine the change in daily heart rate with supplementation from the daily baseline heart rate with 12oz of food colored water. A red food dye will be used to match coloring of supplements.
Change in heart rate from daily baseline with 20g Resync+Collagen | 75-minutes post supplement ingestion
  We will determine the change in daily heart rate with supplementation from the daily baseline heart rate with 1 serving (20g) of Resync+Collagen. This blend contains approximately 17g of collagen, 2 g of Resync, and 1g carbohydrates. Resync+Collagen powder will be mixed with 12oz of water.

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Bloomer, Ph.D., Principal Investigator — Dean of School of Health Studies
Locations (1):
- Center for Nutraceutical and Dietary Supplement Research, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No